CLINICAL TRIAL: NCT02689973
Title: Synergistic Effects of Implementation Intention and Self-efficacy on Behavior Change and Body Fat: a Randomized Controlled Trial of Interventions Promoting Physical Activity
Brief Title: Effects of Self-efficacy, Planning, and Self-efficacy+Planning Interventions on Body Fat Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: University of Zurich (Other); Free University of Berlin (Other); Curtin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N106 036 32/2487
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Adolescent Behavior
Keywords: adolescence; body fat; physical activity; psychosocial intervention; self-efficacy; planning
MeSH Terms: conditions — Adolescent Behavior; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Self-efficacy (Experimental): The self-efficacy intervention protocol included following behavior change techniques (BCT; Michie et al., 2011): barrier identification, prompting focus on past success, and prompting self-talk. Applications of all BCT included references to self-efficacy beliefs. The intervention was integrated into health promotion-nutrition education program (8h). The intervention was applied twice (the baseline and 2-month follow-up).
  Interventions: Behavioral: Self-Efficacy; Behavioral: Education
- Planning (Experimental): The following BCT were included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/coping planning. Applications of all BCT included references to planning.
  The intervention was integrated into health promotion-nutrition education program (8h). The intervention was applied twice (the baseline and 2-month follow-up).
  Interventions: Behavioral: Planning; Behavioral: Education
- Combined planning+self-efficacy (Experimental): This condition included all BCT applied in the planning and self-efficacy arms. The intervention was integrated into health promotion-nutrition education program. The intervention was applied twice (the baseline and 2-month follow-up).
  Interventions: Behavioral: Self-Efficacy; Behavioral: Planning; Behavioral: Education
- Education (Active Comparator): The education group received extended physical activity education program. The physical activity education was integrated into health promotion-nutrition education program.The education program was applied twice (the baseline and 2-month follow-up).
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Self-Efficacy — The introductory part included an abbreviated version of the education materials used in the control group. The self-efficacy materials and forms had four sections: (a) definitions of self-efficacy beliefs, (b) information on the importance of self-efficacy for goal pursuit, (c) recollecting a mastery experience, (d) persuasive statements evoking self-persuasive statements about self-efficacy beliefs. The materials ended with instructions for the following 7 days to recollect self-efficacy enhancing statements every morning. The procedures are based on a self-efficacy intervention by Luszczynska, Tryburcy et al. (2007).
  Group and individual components were included. Setting: secondary and high schools.
  Other Names: Physical Activity Self-Efficacy Enhancement
  Arms: Combined planning+self-efficacy; Self-efficacy
Behavioral: Planning — The introductory part included an abbreviated version of the education materials used in the control group. The planning materials and forms had four sections: (a) information on the importance of planning, including examples of how planning works and what it affects, (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans. The materials ended with instructions for the following 7 days to recollect/redo plans every morning.The procedures are based on a planning intervention by Luszczynska, Sobczyk, et al. (2007).
  Group and individual components were included. Setting: secondary and high schools.
  Other Names: Physical Activity Planning Enhancement
  Arms: Combined planning+self-efficacy; Planning
Behavioral: Education — Participants received a set of educational materials about types of physical activity (PA), PA intensity, exercise calorie expenditure, myths about PA, strength and endurance training, stretching, and general healthy nutrition guidelines. The materials excluded planning and self-efficacy statements.
  The materials ended with instructions for the following 7 days to recollect forms of MVPA every morning.
  Group and individual components were included. Setting: secondary and high schools.
  Other Names: Physical Activity Education

SUMMARY:
This longitudinal experimental study tested the effects of three brief interventions: (1) prompting the formation of plans (or implementation intentions), (2) prompting self-efficacy beliefs, and (3) prompting planning + self-efficacy in adolescents aged 14-18 years relative to an active 'education only' control group.

It was hypothesized that participants assigned to the interventions would exhibit a smaller increase in body fat at 14-month follow-up compared to controls. The study also investigated whether the combined planning + self-efficacy intervention would have larger effects on the main outcome (body fat) than single-component interventions. Second, it was hypothesized that the effects of the intervention conditions on body fat at 14-month follow-up would be mediated by their respective psychological and behavioral constructs: self-efficacy and planning at T2 (Mediator 1), and by moderate-to-vigorous physical activity (MVPA) at T3 (Mediator 2). It was expected that the effects of the interventions including the planning component (i.e., planning intervention and self-efficacy + planning intervention) would be mediated by respective cognitions, i.e. planning, whereas the effects of the interventions including self-efficacy component (i.e., self-efficacy intervention and self-efficacy + planning intervention) would be mediated by self-efficacy. Finally, it was explored whether the effects of the intervention (both direct and indirect effects, via their respective psychological variables and MVPA) on body fat would be moderated by the presence of built PA facilities, located in the proximity of schools.

DETAILED DESCRIPTION:
The experimental procedures were integrated into a health promotion and education program.

Pre-manipulation education: Across the study groups, participants received a common healthy lifestyle education program, focusing on nutrition and physical activity, which was a part of the school curriculum. The combination of nutrition and PA interventions is in line with best practice guidelines for interventions promoting healthy body weight. The education program was delivered by teachers and a group format was used. The groups discussed food composition, safe food handling, food labeling, nutrient needs for age and gender groups, dietary guidelines, and clinical nutrition issues. The program did not include behavior change techniques and was not accompanied by changes in policies.

The intervention conditions were delivered via a combination of printed forms with paper-and-pencil exercises and face-to-face sessions. All experimental conditions included an initial session (completing the forms individually in the groups + face-to-face component) and sets of handouts for three following weeks. The face-to-face component was delivered within three days of completing the initial forms. The initial session was followed by a booster session (group + face-to-face components), delivered at 2-month follow-up. Across the groups, completing the forms (individual component) took approximately 30 minutes and was conducted in classrooms. The face-to-face components took 45-60 minutes and were conducted in the offices of school nurses or school psychologists.

Group intervention component. At the baseline participants completed the intervention materials individually, using self-copy paper; the copies were collected for fidelity analysis and originals were left for participants. The paper-and-pencil materials followed a similar format in four groups in terms of word count, visual format, and the number and length of sections requiring participants filling in the blanks.

Face-to-face intervention component. During the face-to-face component (at the baseline and during the booster sessions) all participants received feedback on their body weight, information regarding their physical activity levels and energy expenditure based on participant's age, gender, body weight, followed by moderate-to-vigorous physical activity recommendations (body mass and body fat measured during the booster session was not recorded). Next, all participants and experimenters jointly reviewed the forms completed during the group component. Adolescents reported included plans and were prompted to provide even more detailed responses to questions included in the forms. Experimenters asked participants to read the content of the form loudly; looked for sections which were incomplete and encouraged adolescents to complete these sections; prompted participants to provide detailed responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents
* Adolescents with chronic conditions but without contraindications for moderate-to-vigorous physical activity

Exclusion Criteria:

* Adolescents who were younger than 14 years old
* Adolescents who declared plans for changing schools during the following year (e.g., due to graduation or moving to another region)
* No parental consent at the baseline
* Existing diseases with contraindications for moderate-to-vigorous physical activity

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1217 (Actual)
Dates: Start 2009-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Luszczynska, PhD, Principal Investigator — University of Social Sciences and Humanities
Locations (1):
- University of Social Sciences and Humanities, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luszczynska A, Schwarzer R, Lippke S, Mazurkiewicz M. Self-efficacy as a moderator of the planning-behaviour relationship in interventions designed to promote physical activity. Psychol Health. 2011 Feb;26(2):151-66. doi: 10.1080/08870446.2011.531571. PMID 21318927
- [Background] Michie S, Ashford S, Sniehotta FF, Dombrowski SU, Bishop A, French DP. A refined taxonomy of behaviour change techniques to help people change their physical activity and healthy eating behaviours: the CALO-RE taxonomy. Psychol Health. 2011 Nov;26(11):1479-98. doi: 10.1080/08870446.2010.540664. Epub 2011 Jun 28. PMID 21678185
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Cleary J, Daniells S, Okely AD, Batterham M, Nicholls J. Predictive validity of four bioelectrical impedance equations in determining percent fat mass in overweight and obese children. J Am Diet Assoc. 2008 Jan;108(1):136-9. doi: 10.1016/j.jada.2007.10.004. PMID 18156000
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Gomez JM, Heitmann BL, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, Schols AM, Pichard C; Composition of the ESPEN Working Group. Bioelectrical impedance analysis--part I: review of principles and methods. Clin Nutr. 2004 Oct;23(5):1226-43. doi: 10.1016/j.clnu.2004.06.004. PMID 15380917
- [Background] Schwarzer R, Luszczynska A, Ziegelmann JP, Scholz U, Lippke S. Social-cognitive predictors of physical exercise adherence: three longitudinal studies in rehabilitation. Health Psychol. 2008 Jan;27(1S):S54-63. doi: 10.1037/0278-6133.27.1(Suppl.).S54. PMID 18248106
- [Background] Luszczynska A, Horodyska K, Zarychta K, Liszewska N, Knoll N, Scholz U. Planning and self-efficacy interventions encouraging replacing energy-dense foods intake with fruit and vegetable: A longitudinal experimental study. Psychol Health. 2016;31(1):40-64. doi: 10.1080/08870446.2015.1070156. Epub 2015 Aug 6. PMID 26160226
- [Background] Luszczynska A, Tryburcy M, Schwarzer R. Improving fruit and vegetable consumption: a self-efficacy intervention compared with a combined self-efficacy and planning intervention. Health Educ Res. 2007 Oct;22(5):630-8. doi: 10.1093/her/cyl133. Epub 2006 Oct 23. PMID 17060349
- [Background] Luszczynska A, Sobczyk A, Abraham C. Planning to lose weight: randomized controlled trial of an implementation intention prompt to enhance weight reduction among overweight and obese women. Health Psychol. 2007 Jul;26(4):507-12. doi: 10.1037/0278-6133.26.4.507. PMID 17605571
- [Result] Luszczynska A, Hagger MS, Banik A, Horodyska K, Knoll N, Scholz U. Self-Efficacy, Planning, or a Combination of Both? A Longitudinal Experimental Study Comparing Effects of Three Interventions on Adolescents' Body Fat. PLoS One. 2016 Jul 13;11(7):e0159125. doi: 10.1371/journal.pone.0159125. eCollection 2016. PMID 27410961

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-efficacy: The self-efficacy intervention protocol included following behavior change techniques (BCT; Michie et al., 2011): barrier identification, prompting focus on past success, prompting self-talk. The intervention was integrated into health promotion-nutrition education program (8h). The intervention was applied twice (the baseline and 2-month follow-up).
  Self-Efficacy: The introductory part included an abbreviated version of the education materials used in the control group. The self-efficacy materials and forms had four sections: (a) definitions of self-efficacy beliefs, (b) information on the importance of self-efficacy for goal pursuit, (c) recollecting a mastery experience, (d) persuasive statements evoking self-persuasive statements about self-efficacy beliefs. The materials ended with instructions for the following 7 days to recollect self-efficacy enhancing statements every morning.
- Planning: The following BCT were included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/coping planning. Applications of all BCT included references to planning.
  The intervention was integrated into health promotion-nutrition education program (8h). The intervention was applied twice (the baseline and 2-month follow-up).
  Planning: The introductory part included an abbreviated version of the education materials used in the control group. The planning materials and forms had four sections: (a) information on the importance of planning, including examples of how planning works and what it affects, (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans. The materials ended with instructions for the following 7 days to recollect/redo plans every morning.The procedures are based on a planning intervention by Luszczynska et al. (2007)
- Combined Planning+Self-efficacy: This condition included all BCT applied in the planning and self-efficacy arms. The intervention was integrated into health promotion-nutrition education program. The intervention was applied twice (the baseline and 2-month follow-up).
  Self-Efficacy: The introductory part included an abbreviated version of the education materials used in the control group. The self-efficacy materials and forms had four sections: (a) definitions of self-efficacy beliefs, (b) information on the importance of self-efficacy for goal pursuit, (c) recollecting a mastery experience, (d) persuasive statements evoking self-persuasive statements about self-efficacy beliefs. The materials ended with instructions for the following 7 days to recollect self-efficacy enhancing statements every morning. The procedures are based on a self-efficacy intervention by Luszczynska, Tryburcy et al. (2007).
  Group and individual components were included. Setting: secondary and high schools.
- Education: The education group received extended physical activity education program. The physical activity education was integrated into health promotion-nutrition education program.The education program was applied twice (the baseline and 2-month follow-up).
  Education: Participants received a set of educational materials about types of physical activity (PA), PA intensity, exercise calorie expenditure, myths about PA, strength and endurance training, stretching, and general healthy nutrition guidelines. The materials excluded planning and self-efficacy statements.
  The materials ended with instructions for the following 7 days to recollect forms of MVPA every morning.
  Group and individual components were included. Setting: secondary and high schools.
Period: Overall Study
Arm/Group | Self-efficacy | Planning | Combined Planning+Self-efficacy | Education
Started | 311 | 270 | 351 | 285
Completed | 257 | 221 | 279 | 232
Not Completed | 54 | 49 | 72 | 53

BASELINE CHARACTERISTICS:
Groups:
- Self-efficacy: The self-efficacy intervention protocol included following behavior change techniques (BCT; Michie et al., 2011): barrier identification, prompting focus on past success, prompting self-talk. Applications of all BCT included references to self-efficacy beliefs. The intervention was integrated into health promotion-nutrition education program (8h). The intervention was applied twice (the baseline and 2-month follow-up).
  Self-Efficacy: The introductory part included an abbreviated version of the education materials used in the control group. The self-efficacy materials and forms had four sections: (a) definitions of self-efficacy beliefs, (b) information on the importance of self-efficacy for goal pursuit, (c) recollecting a mastery experience, (d) persuasive statements evoking self-persuasive statements about self-efficacy beliefs. The materials ended with instructions for the following 7 days to recollect self-efficacy enhancing statements every morning.
- Total: Total of all reporting groups
Arm/Group | Self-efficacy | Planning | Combined Planning+Self-efficacy | Education | Total
Number analyzed (Participants) | 311 | 270 | 351 | 285 | 1217
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.42 (0.84) | 16.49 (0.59) | 16.40 (0.68) | 16.48 (0.63) | 16.44 (0.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 163 | 194 | 166 | 707
  Male | 127 | 107 | 157 | 119 | 510
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 311 | 270 | 351 | 285 | 1217
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 311 | 270 | 351 | 285 | 1217
Categorical BMI: number of participants with overweight/obesity [Count of Participants; unit: Participants] | 53 | 54 | 75 | 48 | 230

OUTCOME MEASURES:

1. Primary Outcome: Body Fat Tissue
Description: bioimpedance (BIA) method (Kyle et al., 2004), which determines the electrical impedance of an electric current through body tissues. Fat tissue was estimated with Schaefer equation for BIA which is considered a reliable index of body fat in adolescent from primarily white backgrounds (Cleary et al., 2008).
Time Frame: Baseline to 14-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of body fat
Groups:
- Self-efficacy: The self-efficacy intervention protocol included following behavior change techniques (BCT; Michie et al., 2011): barrier identification, prompting focus on past success, prompting self-talk. Applications of all BCT included references to self-efficacy beliefs. The intervention was integrated into health promotion-nutrition education program (8h). The intervention was applied twice (the baseline and 2-month follow-up).
  Self-Efficacy: The introductory part included an abbreviated version of the education materials used in the control group. The self-efficacy materials and forms had four sections: (a) definitions of self-efficacy beliefs, (b) information on the importance of self-efficacy for goal pursuit, (c) recollecting a mastery experience, (d) persuasive statements evoking self-persuasive statements about self-efficacy beliefs. The materials ended with instructions for the following 7 days to recollect self-efficacy enhancing statements every morning. The procedures are based
Arm/Group | Self-efficacy | Planning | Combined Planning+Self-efficacy | Education
Number analyzed (Participants) | 311 | 270 | 351 | 285
percentage of body fat
  Body fat at the baseline | 21.12 (7.28) | 21.99 (6.66) | 21.69 (7.16) | 21.81 (6.81)
  Body fat at the 14-month follow-up | 21.93 (6.74) | 22.68 (6.32) | 22.33 (6.75) | 23.41 (5.87)

2. Secondary Outcome: Moderate-to-vigorous Physical Activity (MVPA)
Description: Items from Godin and Shephard's (1985) Leisure-Time Exercise Questionnaire (e.g., 'Considering a 7-day period [a week], how many times on the average do you do the following kinds of exercise for more than 15 minutes during your free time: strenuous exercise [heart beats rapidly], i.e. running, jogging, hockey, soccer, basketball, cross-country skiing, vigorous swimming, vigorous long distance bicycling').
  Number of Items: 2
  Response format: open ended, the participant indicated the number of 15 min blocks of physical activity.
  Scoring: the total (sum) score of 2 items
  Scoring formula: the sum score for the number of minutes of MVPA per week, i.e. individual score = {response to item #1 x 15} + {response to item # 2 x 15})
  The range for the score (i.e. the sum score of 2 items): minimum = 0, maximum = 42
  Interpretation: Higher scores indicate better results (more minutes of MVPA per week)
Time Frame: Baseline to 14-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-efficacy | Planning | Combined Planning+Self-efficacy | Education
Number analyzed (Participants) | 311 | 270 | 351 | 285
units on a scale
  MVPA : baseline | 7.09 (4.56) | 6.81 (3.88) | 7.11 (4.00) | 7.44 (4.17)
  MVPA: 14-month follow-up | 7.18 (3.90) | 7.52 (4.40) | 7.35 (3.44) | 6.83 (3.88)

3. Secondary Outcome: The Use of Physical Activity Planning (the Use of Planning)
Description: Use of physical activity planning was measured with four items (e.g., 'I have my own plan regarding when to engage in exercise of moderate-to-vigorous intensity'; Schwarzer et al., 2008).
  Number of Items: 4
  Response format: Responses ranged from 1 ('definitely not') to 4 ('exactly true').
  Scoring: the total score of 4 items
  Scoring formula: the sum score for the 4 items divided by 4, i.e. {item #1 + item #2 + item #3 + item #4} : 4
  The range for the score (i.e. the sum score of 4 items divided by 4): minimum = 1, maximum = 4
  Interpretation: Higher scores indicate better results (the more frequent use of planning)
Time Frame: Baseline to 2-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-efficacy | Planning | Combined Planning+Self-efficacy | Education
Number analyzed (Participants) | 311 | 270 | 351 | 285
units on a scale
  The use of planning: baseline | 2.68 (0.87) | 2.64 (0.86) | 2.74 (0.86) | 2.66 (0.85)
  The use of planning: 2-month follow-up | 2.60 (0.89) | 2.76 (0.86) | 2.73 (0.88) | 2.66 (0.91)

4. Secondary Outcome: Physical Activity Self-efficacy (PA Self-efficacy)
Description: Physical activity self-efficacy (T1 and T2) was measured with 9 items (e.g., 'I am able to maintain regular MVPA even if I would have to reorganize my daily life'; Luszczynska et al., 2011).
  Number of Items: 9
  Response format: Responses ranged from 1 ('definitely not') to 4 ('exactly true').
  Scoring: the total score of 9 items divided by 9
  Scoring formula: the sum score for the 9 items divided by 9, i.e. {item #1 + item #2 + item #3 + item #4+ item #5 + item #6 + item #7 + item #8 + item #9} : 9
  The range for score (i.e. the sum score of 9 items divided by 4): minimum = 1, maximum = 4
  Interpretation: Higher scores indicate better results (the higher levels of PA self-efficacy)
Time Frame: Baseline to 2-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-efficacy | Planning | Combined Planning+Self-efficacy | Education
Number analyzed (Participants) | 311 | 270 | 351 | 285
units on a scale
  PA self-efficacy: baseline | 2.60 (0.96) | 2.59 (0.91) | 2.70 (0.91) | 2.61 (0.93)
  PA self-efficacy: 2-month follow-up | 2.80 (0.76) | 2.85 (0.72) | 2.82 (0.76) | 2.67 (0.75)

ADVERSE EVENTS:
Time Frame: The baseline and the follow-up (14 months after the baseline)
Description: The experimenters and school headmasters were asked to provide a number of study participants who reported any serious adverse events during the course of the study (if experimenters/headmasters are aware of any such cases). Serious events were defined as absence (over 14 days) or hospitalization (any length) due to any issues which were perceived by a participant as developed due to their physical activity or nutrition behavior. Other adverse events: participants' complains on study protocol.
Arm/Group | Self-efficacy | Planning | Combined Planning+Self-efficacy | Education
All-Cause Mortality (participants affected / at risk) | 0/311 | 0/270 | 0/351 | 0/285
Serious Adverse Events (participants affected / at risk) | 0/311 | 0/270 | 0/351 | 0/285
Other Adverse Events (participants affected / at risk) | 0/311 | 0/270 | 0/351 | 0/285

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes